CLINICAL TRIAL: NCT03223233
Title: Predicting the Severity of Post-cesarean Wound Infections Using Serum Procalcitonin Levels
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, MD,ObGYN, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2016/12.2
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Wound Infection; Cesarean Wound Disruption
MeSH Terms: conditions — Wound Infection | interventions — Procalcitonin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No secondary suture: The participants who developed post-cesarean surgical site infection and follow-up only antibiotic treatment for their wound care.
  Interventions: Other: procalcitonin level
- Secondary suture: The participants who developed post-cesarean surgical site infection and need a secondary suture for their wound care
  Interventions: Other: procalcitonin level

INTERVENTIONS:
Other: procalcitonin level — serum procalcitonin level will be measured in both groups.

SUMMARY:
The serum procalcitonin levels are important during infections and sepsis. The investigators aimed to assess its predictive value in terms of post-cesarean wound infection.

DETAILED DESCRIPTION:
The serum procalcitonin levels are important during infections and sepsis. Recent studies showed that serum procalcitonin levels are more sensitive than serum CRP levels.The investigators aimed to assess its predictive value in terms of post-cesarean wound infection. The serum procalcitonin levels are aimed to measure in participants who had cesarean section and developed surgical site infection. The investigators aimed to compare the serum procalcitonin levels between the patients who need secondary suture and the patients who did not need secondary suture.

ELIGIBILITY:
Inclusion Criteria:

* who developed surgical site infection after their cesarean sections.
* 18-40 years old

Exclusion Criteria:

* history of chorioamnionitis and premature rupture of membranes
* urinary tract infections
* any infectious condition other than surgical site infection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients who underwent cesarean section
Study Population: The participants are post-cesarean patients who developed surgical site infections.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-10-08 (Actual)

PRIMARY OUTCOMES:
Serum procalcitonin levels in participants who developed wound infection after cesarean sections | 5 months
  Serum procalcitonin levels will be measured in participants who will develop post-cesarean wound site infections. The serum procalcitonin levels will be compared in subgroups who need secondary suture and those who don't require suturing

CONTACTS AND LOCATIONS:
Overall Officials: Alev Atis, MD,ObGyn, Study Director — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni SSRTH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wacker C, Prkno A, Brunkhorst FM, Schlattmann P. Procalcitonin as a diagnostic marker for sepsis: a systematic review and meta-analysis. Lancet Infect Dis. 2013 May;13(5):426-35. doi: 10.1016/S1473-3099(12)70323-7. Epub 2013 Feb 1. PMID 23375419
- [Background] Takakura Y, Hinoi T, Egi H, Shimomura M, Adachi T, Saito Y, Tanimine N, Miguchi M, Ohdan H. Procalcitonin as a predictive marker for surgical site infection in elective colorectal cancer surgery. Langenbecks Arch Surg. 2013 Aug;398(6):833-9. doi: 10.1007/s00423-013-1095-0. Epub 2013 Jun 20. PMID 23784676
- [Result] Erenel H, Yilmaz N, Oncul M, Acikgoz AS, Karatas S, Ayhan I, Aslan B, Tuten A. Usefulness of Serum Procalcitonin Levels in Predicting Tubo-Ovarian Abscess in Patients with Acute Pelvic Inflammatory Disease. Gynecol Obstet Invest. 2017;82(3):262-266. doi: 10.1159/000449161. Epub 2016 Sep 3. PMID 27592364
- [Derived] Aslan Cetin B, Aydogan Mathyk B, Koroglu N, Temel Yuksel I, Konal M, Erenel H, Atis Aydin A. Serum procalcitonin levels in incisional surgical site infections requiring a secondary suture after cesarean sections. J Matern Fetal Neonatal Med. 2019 Dec;32(24):4108-4113. doi: 10.1080/14767058.2018.1481949. Epub 2018 Jun 20. PMID 29804483